CLINICAL TRIAL: NCT04865783
Title: Cryospray to Reduce Pain During Venous Cannulation - Randomized Placebo-controlled Study
Brief Title: Cryospray to Reduce Pain During Venous Cannulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: SHS-BI-4a-2021
Record Dates: First submitted 2021-04-28; First posted 2021-04-29 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Catheterization; Anesthetics, Intravenous; Elective Surgical Procedures
Keywords: cryospray

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Before elective surgery, all patients will have an intravenous line placed before induction of anaesthesia. Patients will be blinded to whether cryospray or placebo is used. Two anaesthesia trained persons (nurse/doctors) will perform the procedure. One person will randomize and apply the randomized spray and the other person will be blinded to the randomized treatment. The anesthesiologist performing the puncture but blinded for randomization will fill out a questionnaire
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryospray (Active Comparator): Cryospray will be sprayed from a distance of 20-30 cm to the back of one hand.
  Interventions: Procedure: Cryospray
- Placebo (Placebo Comparator): A saline solution will be sprayed from a distance of 20-30 cm to the back of the hand.
  Interventions: Procedure: Saline spray

INTERVENTIONS:
Procedure: Saline spray — The saline spray will be applied twice for 1-2 seconds.
  Arms: Placebo
Procedure: Cryospray — The cryospray will be applied twice for 1-2 seconds.
  Arms: Cryospray

SUMMARY:
This trial aims to evaluate if cryospray can reduce pain during intravenous cannulation in elective surgery compared to a placebo spray.

DETAILED DESCRIPTION:
Venous cannulation is a common practice in the health care system. Before any procedure, intravenous access is always placed before induction of any anaesthesia. For many patients placement of a venous catheter is associated with pain and discomfort. Any quick and easy reduction in pain during the procedure is important for patients. Cryospray has been described as an easy-to-use supplement of analgesia to alleviate pain during intravenous access. Cryospray has been shown to reduce pain in venous cannulation in the emergency setting but not in the elective setting. A search in the literature reveals 2 recent metanalyses reporting 8 included trials and 11 included trials, respectively. Both metanalyses call for further research in relation to patients' satisfaction. By randomizing patients to either cryospray or placebo before venous cannulation, we hypothesize that cryospray reduces pain during venous cannulation compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older and able to give consent

Exclusion Criteria:

* Unable to give consent
* Infection
* coloring or bruises at the puncture site (use of corticosteroid etc).
* No vein signs visible after application of vein stasis.
* Allergy to coolant spray.
* Contraindication for vein stasis or vein cannulation (ex Raynauds disease etc).
* Has participated earlier in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Patients reported pain from the puncture site | immediately after completion of vein canulation
  After vein puncture is completed patients is asked on a scale from 0-10 to indicate pain during vein canulation (zero no pain, 10 worst possible pain)

SECONDARY OUTCOMES:
Difficulty in placement of intravenous line | immediately after completion of vein canulation
  After vein puncture is completed the operator is asked to the difficulty in placement of the venous line (0-10, zero very easy and ten very difficult).
Number of successful placements of venous line at first attempt | immediately after completion of vein canulation
  After vein puncture is completed it is indicated wether or not it was successful in first attempt.

OTHER OUTCOMES:
Discomfort from puncture site at discharge from recovery | up to 24 hours after discharge from recovery room
  After discharge from the recovery room patients is asked for any discomfort at the puncture site. If yes: pain, numbness, burning or cold feeling. All positive values rated on the numeric rating scale (0-10).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Strøm, Principal Investigator — University Hospital of Southern Denmark
Locations (1):
- Sygehus Soenderjylland, Aabenraa, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mace SE. Prospective, randomized, double-blind controlled trial comparing vapocoolant spray vs placebo spray in adults undergoing venipuncture. Am J Emerg Med. 2016 May;34(5):798-804. doi: 10.1016/j.ajem.2016.01.002. Epub 2016 Jan 7. PMID 26979261
- [Background] Griffith RJ, Jordan V, Herd D, Reed PW, Dalziel SR. Vapocoolants (cold spray) for pain treatment during intravenous cannulation. Cochrane Database Syst Rev. 2016 Apr 26;4(4):CD009484. doi: 10.1002/14651858.CD009484.pub2. PMID 27113639
- [Background] Zhu Y, Peng X, Wang S, Chen W, Liu C, Guo B, Zhao L, Gao Y, Wang K, Lou F. Vapocoolant spray versus placebo spray/no treatment for reducing pain from intravenous cannulation: A meta-analysis of randomized controlled trials. Am J Emerg Med. 2018 Nov;36(11):2085-2092. doi: 10.1016/j.ajem.2018.03.068. Epub 2018 Mar 27. PMID 30253890
- [Derived] Pedersen JB, Martensen A, Funder P, Bakke SA, Bhavsar RP, Strom T. Cryospray reduces pain during venous cannulation in elective surgery patients: a randomized placebo-controlled study. BMC Anesthesiol. 2024 Dec 19;24(1):466. doi: 10.1186/s12871-024-02858-2. PMID 39702029